CLINICAL TRIAL: NCT01398163
Title: A f-MRI STUDY OF AFFECTIVE CHANGES ASSOCIATED WITH FOUR WEEKS CONSUMPTION OF A FERMENTED DAIRY PRODUCT IN HEALTHY WOMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU271
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Adult Women
Keywords: probiotics; digestive well-being; fMRI; brain-gut axis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 = Tested product (Experimental)
  Interventions: Other: 1-Fermented Dairy Product (test)
- 2 = Control product (Active Comparator)
  Interventions: Other: 2-Milk-based non-fermented dairy product(control)
- 3 = No product (No Intervention)

INTERVENTIONS:
Other: 1-Fermented Dairy Product (test) — Arm 1 - Intervention 1 (probiotics)
  Arms: 1 = Tested product
Other: 2-Milk-based non-fermented dairy product(control) — Arm 2 - Intervention 2 (control)
  Arms: 2 = Control product

SUMMARY:
The purpose of this study is to evaluate the effect of a commercially available fermented dairy product containing probiotics (4 weeks, twice a day) on the brain activity within specific neural circuits regulating the subjective experience of emotional valence and digestive well-being.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, right-handed, aged from 18 to 60 years
* Subject of normal body weight or with overweight i.e. not obese (body mass index between 18 and 30 kg/m2).
* For fertile women, complying with one of the other medically approved methods of contraception

Exclusion Criteria:

* Subject with any current psychiatric or eating or suicidal attempt disorder, or history of such disorder.
* Subject with any history of chronic GI disorder or disease.
* Subject with any significant active or prior metabolic disorder or disease.
* Subject with any use of probiotic supplements or antibiotics in the previous month.
* Subject with current use of any medications with potential central nervous system effects (antidepressants, anxiolytics, opiate pain medications...).
* Subject with allergy or hypersensitivity to milk proteins or lactose intolerance or immunodeficiency
* Subjects with claustrophobia or other condition (such as metallic implants) that would preclude MRI scanning

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA - University, Los Angeles, California, United States